CLINICAL TRIAL: NCT04192955
Title: Evaluating Oral Peri-operative Acetylsalicylic Acid in Subjects Undergoing Endovascular Coiling-only of Unruptured Brain Aneurysms(EVOLVE): A Phase 3 Multicenter Randomized Study
Brief Title: Evaluating Oral Peri-operative Acetylsalicylic Acid in Subjects Undergoing Endovascular Coiling-only of Unruptured Brain Aneurysms
Acronym: EVOLVE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Version 2.0
Record Dates: First submitted 2019-11-28; First posted 2019-12-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Unruptured Cerebral Aneurysm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Acetylsalicylic acid (ASA) will be given orally at a dose of 324 mg to be taken daily starting 3 days prior to the planned coiling procedure day, on the procedure day, and for one-day post-procedure.
  Interventions: Drug: Acetyl Salicylate
- Control (Placebo Comparator): Lactose100-mg tablets to be taken daily starting 3 days prior to the planned coiling procedure day, on the procedure day, and for one-day post-procedure.
  Interventions: Drug: Acetyl Salicylate

INTERVENTIONS:
Drug: Acetyl Salicylate — Tablets

SUMMARY:
This trial is a is a prospective, randomized (1:1) placebo-controlled, clinical trial with blinded endpoint assessment of 440 participants with unruptured brain aneurysm planned for endovascular treatment using coiling-only approach (primary coiling or using balloon-assistance but not stenting) to test if oral acetylsalicylic acid (325 mg/ day for a total of 5 days) is superior placebo in preventing clinical and silent strokes. The primary outcome is a clinical or silent stroke at the time of discharge assessed by clinical examination and MRI brain. Participants will return to the clinic or be contacted by phone for the end of study procedures on Day 90 to collect functional outcome data.

DETAILED DESCRIPTION:
Endovascular aneurysm treatment has become the mainstay of treatment of unruptured brain aneurysms. Since the introduction of Guglielmi detachable coils in the late 1980s, thousands of procedures are performed annually worldwide. The expanding endovascular armamentarium with the use of balloon-assisted coiling, stents (either in stent-assisted coiling or flow-diversion), and unassisted coiling-only procedures made it possible to treat aneurysms of almost all intracranial locations, shapes, and sizes.

Thromboembolic complications are potential adverse events whenever catheters are introduced into the intracranial arteries. Diagnostic and interventional neurological procedures, such as diagnostic and therapeutic cerebral angiograms may lead to ischemic strokes of varying frequency and severity. Luckily, most of the thromboembolic events do not cause a clinical stroke. Instead, tiny infarction signals are seen on Diffusion-weighted magnetic resonance imaging (DWI MRI) of the brain without neurological signs or symptoms. These are often labelled as silent (or covert) strokes. These imaging surrogates have been used to compare the safety and efficacy of various endovascular procedures and techniques. In a Canadian cohort, heparin bolus during aneurysm coiling was associated with significantly less DWI load on post-coiling MRI. This supports the notion that most of these lesions are caused by thrombi, as opposed to bubbles.

There is limited direction from available guidelines regarding the use of anticoagulation or antiplatelet agents to prevent thromboembolic complications associated with endovascular treatment of brain aneurysms. This resulted in huge variability of the protocols used for anticoagulation and antiplatelet therapies before, during and after coil embolization of brain aneurysms. Most of the current practices are extrapolated from coronary literature.

Platelet inhibition is an effective strategy to minimize the rate of thromboembolism. Antiplatelet treatment has been routinely used before coronary angioplasty to reduce the risk of thromboembolic events. The different action of ASA from that of anticoagulants gives it an additive effect to heparin alone in neuro-interventional procedures. This notion is supported by observations from multiple retrospective and prospective studies.

We will perform a prospective, randomized (1:1) placebo-controlled, clinical trial with blinded endpoint assessment of 440 participants with unruptured brain aneurysm planned for endovascular treatment using coiling-only approach (primary coiling or using balloon-assistance but not stenting) to test if oral acetylsalicylic acid (325 mg/ day for a total of 5 days: 3 days prior and two days after and including the coiling procedure day) is superior placebo in preventing clinical and silent strokes. The primary outcome is a clinical or silent stroke at the time of discharge assessed by clinical examination and MRI brain.

ELIGIBILITY:
Inclusion Criteria:

* Unruptured intracranial aneurysm suitable for coiling-only (primary coiling or balloon-assisted) as a primary treatment.
* Functionally independent at baseline (modified Rankin scale <3).
* Informed consent and availability of the subject for the entire study period.

Exclusion Criteria:

1. Planned complex aneurysm treatment including use of any device that requires post-operative antiplatelet therapy (stent-assisted coiling or flow-diverter device), or endovascular vessel sacrifice.
2. Dissecting or mycotic brain aneurysm.
3. Any ongoing ischemic symptoms such as transient ischemic attacks, minor strokes, or stroke-in-evolution within 2 weeks before randomization.
4. Allergy or contraindication to ASA.
5. Unable to take study drug orally for any reason.
6. Subjects already taking single or dual antiplatelet, warfarin, or any of the non-Vitamin K antagonist oral anticoagulants.
7. Subjects unable to undergo MRI imaging for any reason (e.g., severe claustrophobia or presence of metals).
8. Any other medical condition that the site investigator deems would put the subject at excessive risk by participation in the study (e.g. active bleeding, symptomatic peptic ulcer disease, liver or kidney failure, thrombocytopenia or coagulopathy) or an expected life expectancy less than one year, or that would result in an inability to collect radiological outcomes and clinical outcomes at 90 days.
9. Pregnancy or breastfeeding.
10. Prior enrollment in EVOLVE trial for another aneurysm.
11. Participation in another clinical trial of an investigational drug, device or procedure if the subject received the trial drug, device or procedure in the preceding 30 days from the anticipated coiling date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical or silent stroke | within 2-4 days of completion of the coiling procedure
  Incidence of embolic strokes (clinically or on DWI-MRI)

SECONDARY OUTCOMES:
Symptomatic stroke | Day 90 following coiling.
  Clinical thromboembolic events
Death rate | within 90 days following coiling
Peri-operative hemorrhagic complication | within 90 days following coiling
  intracranial hemorrhage, retroperitoneal hematoma, upper or lower gastrointestinal bleeding, or any bleeding stratified as major according to thrombolysis in myocardial infarction (TIMI) definition.
Count of new DWI lesions on post-coiling MRI | within 2-4 days of completion of the coiling procedure
Total volume of new DWI lesions on post-coiling MRI | within 2-4 days of completion of the coiling procedure
Frequency of large (> 10 cc volume) strokes on DWI MRI | within 2-4 days of completion of the coiling procedure
Incidence of cognitive decline on Montreal Cognitive Assessment (MoCA) from baseline to discharge. | within 2-4 days of completion of the coiling procedure
Incidence of visible thrombus formation during the coiling procedure | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Almekhlafi, MD MSc FRCPC, Principal Investigator — University of Calgary; Mayank Goyal, MD PhD FRCPC, Principal Investigator — University of Calgary; Linda Andersen, PhD, Study Director — University of Calgary; Craig Doram, PEng, Study Director — University of Calgary
Locations (9):
- Canada (8):
  - Foothills Medical Center, Calgary, Alberta
  - U of Alberta, Edmonton, Alberta
  - Dalhousie University, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Toronto St Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Centre Hospitalier Régional Universitaire de Tours, Tours, Centre-Val de Loire, France

IPD SHARING:
Plan to Share IPD: No